CLINICAL TRIAL: NCT00797992
Title: Bevacizumab Intravitreal for Myopic Choroidal Neovascularization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JN-05-2008-AR
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Myopic Choroidal Neovascularization
Keywords: Bevacizumab; Myopia; Complications; Neovascularization; OCT
MeSH Terms: conditions — Myopia; Neovascularization, Pathologic | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Myopic eyes with retinal neovascularization
  Interventions: Drug: Injection

INTERVENTIONS:
Drug: Injection — Intravitreal injection of 1.25 mg bevacizumab

SUMMARY:
To evaluate the clinical results of anti-VEGF intra-vitreal injections (IVT) in CNV secondary to pathologic myopia (PM-CNV).

DETAILED DESCRIPTION:
Nineteen consecutive patients (19 eyes) with subfoveal PM-CNV, 18 of whom had been unsuccessfully treated with Visudyne PDT, were treated with IVT of 1.25 mg bevacizumab or 0.5mg ranibizumab. ETDRS best corrected visual acuity, macular thickness on OCT scans, and angiographic features were recorded and evaluated. The aspect of OCT scans passing across the PM-CNV was also analyzed. IVTs were repeated only in case of persistent angiographic leakage and if OCT scans showed retinal thickening or edema and serous retinal detachment. The follow-up period was at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Myopic CNVM,

Exclusion Criteria:

* Patients with poor compliance
* Patients with uncontrolled diabetes and hypertension or any other medical condition that increase the risk of complications like recent history of Stroke or myocardial infraction (< one year). (Physician clearance was obtained for all patients).
* Age related macular degeneration with Juxtafoveal and Subfoveal CNVM: Recurrent CNVM following PDT and TTT with IVTA. Patient who could not afford PDT, Macugen or Lucentis which is FDA approved.
* Patients who had undergone major surgery 28 days before, were excluded from the study and it was also suspended prior to elective surgery.
* Refractory macular oedema due to vein occlusion, Pseudophakia, Clinically significant macular oedema (CSME) etc. that affects vision and does not respond adequately to usual treatment methods.
* Proliferative diabetic retinopathy, non-resolving vitreous haemorrhage with PDR.
* Idiopathic CNVM, Inflammatory CNVM and other conditions associated with CNVM.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao J Nassaralla, PhD, Study Chair — Instituto de Olhos de Goiania
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil